CLINICAL TRIAL: NCT05103943
Title: Amyloidosis TTR Flow Reserve Evaluation
Acronym: AMYTRE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHRO-2021-05
Record Dates: First submitted 2021-09-30; First posted 2021-11-02 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Amyloid Cardiomyopathy
Keywords: Tafamidis
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPECT MPI (myocardial perfusion imaging) Group (Experimental): the SPECT MPI protocol will be modified to evaluated MBF and MFR. This modification will result in no added radiation; the radiopharmaceutical dose will still be the same compared to a standard MPI protocol.
  Interventions: Other: SPECT MPI

INTERVENTIONS:
Other: SPECT MPI — SPECT MPI including dynamic acquisitions for stress, rest MBF and MFR

SUMMARY:
Anginal symptoms and signs of ischemia have been reported in some patients with cardiac amyloidosis (TTR) without obstructive epicardial coronary artery disease (CAD).

It was found that coronary microvascular dysfunction was highly prevalent in subjects with cardiac amyloidosis, even in the absence of epicardial CAD. The investigators found lower stress and rest myocardial blood flow (MBF) and lower myocardial flow reserve (MFR) in their cardiac PET (Positron emission tomography) study (13N), including 21 patients.

The advances in SPECT technology including cadmium zinc telluride (CZT) detectors allow to evaluate the MBF and MFR estimation by SPECT as shown in both experimental animal models and also in clinical studies with comparison to PET.

SPECT is more widely available than cardiac PET.

DETAILED DESCRIPTION:
Anginal symptoms and signs of ischemia have been reported in some patients with cardiac amyloidosis (TTR) without obstructive epicardial coronary artery disease (CAD).

It was found that coronary microvascular dysfunction was highly prevalent in subjects with cardiac amyloidosis, even in the absence of epicardial CAD. The investigators found lower stress and rest myocardial blood flow (MBF) and lower myocardial flow reserve (MFR) in their cardiac PET (Positron emission tomography) study (13N), including 21 patients.

The advances in SPECT technology including cadmium zinc telluride (CZT) detectors allow to evaluate the MBF and MFR estimation by SPECT as shown in both experimental animal models and also in clinical studies with comparison to PET.

SPECT is more widely available than cardiac PET. Thus, the investigators would like:

1. to confirm the results of Dorbala et al using SPECT, and
2. to go further with evaluation of the effect of Tafamidis on microvascular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 90 years
* Understanding and speaking French
* With TTR amyloid cardiomyopathy (ATTRxt or ATTRm) confirmed by the association of heart failure, syncope or bradyarrhythmia, with electrocardiogram and/or magnetic resonance imaging (CMR) suggesting/indicating cardiac amyloid, grade 2 or 3 99mTc- PYP or bone scintigraphy and negative biological findings (i.e. serum immunofixation, urine immunofixation, serum free light chain assay); or, if one of those criteria is not met, presence of amyloid deposits on analysis of biopsy specimens obtained from cardiac and non-cardiac sites (17-19),
* Intention to treat (Tafamidis)

Exclusion Criteria:

* Heart failure not due to transthyretin amyloid cardiomyopathy;
* New York Heart Association (NYHA) class IV heart failure.
* The presence of light-chain amyloidosis;
* A history of liver or heart transplantation;
* An estimated glomerular filtration rate lower than 25 mL per minute per 1.73 m2 of bodysurface area (Cockcroft).
* Liver transaminase levels exceeding two times the upper limit of the normal range;
* Severe malnutrition as defined by a modified body-mass index (mBMI) of less than 600, calculated as the serum albumin level in grams per litter multiplied by the conventional BMI (the weight in kilograms divided by the square of the height in meters);
* Patients receiving concurrent treatment with nonsteroidal anti-inflammatory drugs, tauroursodeoxycholate, doxycycline, calcium-channel blockers, or digitalis;
* Previous treatment with tafamidis or patisaran;
* Ticagrelor treatment
* Previous CAD, severe epicardial stenosis with revascularization or ticagrelor treatment, coronary artery bypass grafting, myocardial infarction;
* Contra-indications to pharmacological stress testing MPI: severe hypotension (< 90 mmHg of Systolic arterial pressure), atrioventricular block 2nd or 3rd grade, carotid stenosis (unilateral >70%, bilateral >50%);
* Pregnancy
* Breastfeeding
* Protected adults
* Other study participation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2026-12-11 (Estimated); Study Completion 2026-12-11 (Estimated)

PRIMARY OUTCOMES:
Difference of Stress and Rest Myocardial Blood Flow | Month 24
  Difference of Stress and Rest Myocardial Blood Flow (mL/min/g) at baseline and after 24 months of treatments, assessed by dynamic SPECT (regional and global left ventricle measurements)
ratio of Stress Myocardial Blood Flow/ Rest Myocardial Blood Flow | Month 24
  Difference of Myocardial Flow Reserve (ie ratio of Stress Myocardial Blood Flow/ Rest Myocardial Blood Flow) at baseline and after 24 months of treatments, assessed by dynamic SPECT (regional and global left ventricle measurements)

SECONDARY OUTCOMES:
Number or participants with stress reduction | baseline
  Stress assessed by dynamic SPECT (regional and global left ventricle measurements), in comparison to "normal" values
Number or participants with rest MBF (myocardial blood flow) reduction | baseline
  Rest Myocardial Blood Flow (mL/min/g) assessed by dynamic SPECT (regional and global left ventricle measurements), in comparison to "normal" values
ratio of Stress Myocardial Blood Flow/ Rest Myocardial Blood Flow | Baseline
  Myocardial Flow Reserve (ie ratio of Stress Myocardial Blood Flow/ Rest Myocardial Blood Flow) assessed by dynamic SPECT (regional and global left ventricle measurements) in comparison to "normal" values

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu BAILLY, Dr, Principal Investigator — CHU Orléans
Locations (4):
- France (4):
  - CHU d'ANGERS, Angers
  - CHU Caen, Caen
  - CHU Orleans, Orléans
  - CHRU de TOURS, Tours

REFERENCES:
- [Background] Dorbala S, Vangala D, Bruyere J Jr, Quarta C, Kruger J, Padera R, Foster C, Hanley M, Di Carli MF, Falk R. Coronary microvascular dysfunction is related to abnormalities in myocardial structure and function in cardiac amyloidosis. JACC Heart Fail. 2014 Aug;2(4):358-67. doi: 10.1016/j.jchf.2014.03.009. Epub 2014 Jul 9. PMID 25023822
- [Background] Maurer MS, Schwartz JH, Gundapaneni B, Elliott PM, Merlini G, Waddington-Cruz M, Kristen AV, Grogan M, Witteles R, Damy T, Drachman BM, Shah SJ, Hanna M, Judge DP, Barsdorf AI, Huber P, Patterson TA, Riley S, Schumacher J, Stewart M, Sultan MB, Rapezzi C; ATTR-ACT Study Investigators. Tafamidis Treatment for Patients with Transthyretin Amyloid Cardiomyopathy. N Engl J Med. 2018 Sep 13;379(11):1007-1016. doi: 10.1056/NEJMoa1805689. Epub 2018 Aug 27. PMID 30145929
- [Background] Al Suwaidi J, Velianou JL, Gertz MA, Cannon RO 3rd, Higano ST, Holmes DR Jr, Lerman A. Systemic amyloidosis presenting with angina pectoris. Ann Intern Med. 1999 Dec 7;131(11):838-41. doi: 10.7326/0003-4819-131-11-199912070-00007. PMID 10610629
- [Background] Ogawa H, Mizuno Y, Ohkawara S, Tsujita K, Ando Y, Yoshinaga M, Yasue H. Cardiac amyloidosis presenting as microvascular angina--a case report. Angiology. 2001 Apr;52(4):273-8. doi: 10.1177/000331970105200407. PMID 11330510
- [Background] Whitaker DC, Tungekar MF, Dussek JE. Angina with a normal coronary angiogram caused by amyloidosis. Heart. 2004 Sep;90(9):e54. doi: 10.1136/hrt.2004.038984. PMID 15310723
- [Background] Nam MC, Nel K, Senior R, Greaves K. Abnormal Myocardial Blood Flow Reserve Observed in Cardiac Amyloidosis. J Cardiovasc Ultrasound. 2016 Mar;24(1):64-7. doi: 10.4250/jcu.2016.24.1.64. Epub 2016 Mar 24. PMID 27081447
- [Derived] Vancon B, Bisson A, Courtehoux M, Bernard A, Bailly M. A study protocol for an observational cohort investigating cardiac transthyretin amyloidosis flow reserve before and after Tafamidis treatment: The AMYTRE study. Front Med (Lausanne). 2022 Aug 23;9:978293. doi: 10.3389/fmed.2022.978293. eCollection 2022. PMID 36082269